CLINICAL TRIAL: NCT00723008
Title: Effect of Cranial Electrotherapy Stimulation on PTSD in Burned Outpatients
Brief Title: Cranial Electrotherapy Stimulation in Burned Patients
Acronym: CES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H-07-024
Record Dates: First submitted 2007-12-25; First posted 2008-07-28 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-02

CONDITIONS: Post Traumatic Stress Disorders; Burns
Keywords: anxiety; insomnia; pain; Alpha Stim; Cranial electrotherapy stimulation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Burns; Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Upon randomization, a double blinded Alpha Stim 100 device preset to the lowest effective setting (1/6) will be applied to the earlobes of the subject for one hour per day for 5 days per week for 4 weeks; after the blinded period is completed the patient will wear a different Alpha Stim device that has not been blinded for one hour per day for 5 days per week for 4 weeks, with settings at the patient's preference (1 to 6/6). Report of pain, anxiety will be assessed before and after each daily session during the 8 week period.
  Interventions: Device: Alpha Stim 100 (Cranial Electrotherapy Stimulation)
- B (Experimental): Upon randomization, a double blinded Alpha Stim 100 device preset to no stimulation (0/6)will be applied to the earlobes of the subject for one hour per day for 5 days per week for 4 weeks; after the blinded period is completed the patient will wear a different Alpha Stim device that has not been blinded for one hour per day for 5 days per week for 4 weeks, with settings at the patient's preference (1 to 6/6). Report of pain, anxiety will be assessed before and after each daily session during the 8 week period.
  Interventions: Device: Alpha Stim 100 (Cranial Electrotherapy Stimulation)

INTERVENTIONS:
Device: Alpha Stim 100 (Cranial Electrotherapy Stimulation) — cranial electrical stimulation 100 microamps
  Other Names: Alpha Stim 100- Electromedical Products International, Inc

SUMMARY:
To find out if Cranial Electrotherapy Stimulation is a useful treatment for people who have been burned and have Post Traumatic Stress Disorder. CES may be helpful in giving relief to some or all of those symptoms.

DETAILED DESCRIPTION:
The purpose of this research study is to systematically determine if CES therapy is effective in managing post traumatic stress disorder (PTSD) in the burn patient. Cranial Electrotherapy Stimulation (CES) is the delivery of low-level electrical stimulation across the head, delivered with ear lobe electrode clips or self-adhesive electrode pads. CES in the current form has been used for the past 30 years to successfully treat anxiety, depression, insomnia and pain in a variety of patient populations. This FDA approved medical device is non-invasive and has no reported significant side effects. It will be used on patients undergoing outpatient rehabilitation in our burn center.

ELIGIBILITY:
Inclusion Criteria:

* burned patients requiring outpatient physical or occupational therapy in the USAISR Burn Rehabilitation Gym or Center for the Intrepid
* Able to read and speak English
* Between ages of 18-65 years
* Screen positive (score greater than 44) on the PCL-M/C instruments

Exclusion Criteria:

* pregnant patients
* patients with implantable pacemakers or electronic stimulators
* patients scoring below 44 on the PCL-M/C instrument
* patients who previously used CES therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-05; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Gaylord, RN, MSN, PhD, Principal Investigator — United States Army Institute of Surgical Research
Locations (1):
- USAISR, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Schroeder MJ, Barr RE. Quantitative analysis of the electroencephalogram during cranial electrotherapy stimulation. Clin Neurophysiol. 2001 Nov;112(11):2075-83. doi: 10.1016/s1388-2457(01)00657-5. PMID 11682346

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Military service members who received outpatient rehabilitation through the US Army Institute of Surgical research (USAISR) were enrolled September 12, 2007-January 9,2009.
Groups:
- A: Active/Unblinded: Upon randomization, a double blinded Alpha Stim 100 device preset to the lowest effective setting (1/6) will be applied to the earlobes of the subject for one hour per day for 5 days per week for 4 weeks; after the blinded period is completed the patient will wear a different Alpha Stim device that has not been blinded for one hour per day for 5 days per week for 4 weeks, with settings at the patient's preference (1 to 6/6). Report of pain, anxiety will be assessed before and after each daily session during the 8 week period.
  Alpha Stim 100 (Cranial Electrotherapy Stimulation) : cranial electrical stimulation 100 microamps
- B: Sham/Unblinded: Upon randomization, a double blinded Alpha Stim 100 device preset to no stimulation (0/6)will be applied to the earlobes of the subject for one hour per day for 5 days per week for 4 weeks; after the blinded period is completed the patient will wear a different Alpha Stim device that has not been blinded for one hour per day for 5 days per week for 4 weeks, with settings at the patient's preference (1 to 6/6). Report of pain, anxiety will be assessed before and after each daily session during the 8 week period.
  Alpha Stim 100 (Cranial Electrotherapy Stimulation) : cranial electrical stimulation 100 microamps
Period: Enrollment
Arm/Group | A: Active/Unblinded | B: Sham/Unblinded
Started | 11 | 9
Completed | 10 | 9
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: 4-Week Double Blinded
Arm/Group | A: Active/Unblinded | B: Sham/Unblinded
Started | 10 | 9
Completed | 5 | 4
Not Completed | 5 | 5
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 4 | 3
Period: 4-Week Unblinded Treatment
Arm/Group | A: Active/Unblinded | B: Sham/Unblinded
Started | 5 | 4
Completed | 4 | 3
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Active/Unblinded | B: Sham/Unblinded | Total
Number analyzed (Participants) | 11 | 9 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 26.3 (4.9) | 27.3 (4.9) | 26.8 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 9 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 5 | 8 | 13
  African American | 3 | 0 | 3
  Hispanic | 3 | 0 | 3
  Other, not specified | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Post-Traumatic Stress Questionnaire-Military (PCL-M) Score
Description: Subjects were asked to complete questionnaire three times during the course of study. Questions addressed symptoms associated with Post Traumatic Stress Disorder(PTSD). Scores can range from 17 to 85. A score >31 was used to identify symptomatic subjects and was therefore required at baseline for study enrollment.
Time Frame: Baseline, Week 4, Week 8
Population: All active subjects
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | A: Active/Unblinded | B: Sham/Unblinded
Number analyzed (Participants) | 11 | 9
Score
  Baseline | 53.8 (16.4) | 56.7 (9.6)
  Week 4 | 48.8 (15.3) | 50.4 (17.1)
  Week 8 | 55.5 (14.8) | 44.7 (2.1)

2. Primary Outcome: Mean Center for Epidemiological Studies-Depression Scale (CES-D) Score
Description: This 20-item questionnaire measures depressive symptoms. Scores can range from 0-60, with scores greater than 16 indicating need for further evaluation due to possible Major Depression.
Time Frame: Baseline, 4 Weeks, 8 Weeks
Population: One A:Active/Unblinded subject was removed from analysis due to a 31-point outlying score. All other subjects who remained in study at each given period were analyzed. Therefore, the number of subjects examined decreased at each interval.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | A: Active/Unblinded | B: Sham/Unblinded
Number analyzed (Participants) | 10 | 9
Score
  Baseline | 28.8 (8.9) | 30.6 (9.9)
  Week 4 | 27.5 (8.2) | 24.5 (13.0)
  Week 8 | 36.3 (4.5) | 21.7 (9.8)

3. Primary Outcome: Mean Brief Profile of Mood States (BPOMS) Score
Description: BPOMS is a tool used to qualitatively measure anxiety. Subjects were asked to evaluate 30 feelings that they may have had over the past week. Stress-associated feelings are scored on a 5-point Likert scale from 0 (not at all)to 4 (extremely). Six of the feelings listed on the questionnaire are not associated with anxiety and therefore are not scored. Total scores range from 0-96, with higher scores indicating greater tension and anxiety.
Time Frame: Baseline, Week 4, Week 8
Population: One A:Active/Unblinded subject was removed from analysis due to a 39-point outlying score. All other subjects who remained in study at each given period were analyzed. Therefore, the number of subjects examined decreased at each interval.
Measure: Mean (Standard Deviation); unit: Brief POMS Score
Arm/Group | A: Active/Unblinded | B: Sham/Unblinded
Number analyzed (Participants) | 10 | 9
Brief POMS Score
  Baseline | 50.2 (21.7) | 55.9 (15.4)
  Week 4 | 42.3 (21.9) | 50.3 (10.3)
  Week 8 | 51.0 (11.5) | 41.0 (9.9)

4. Primary Outcome: Mean Visual Analogue Scale of Pain (VAS-P) Before and After Cranial Electrotherapy Stimulation (CES).
Description: Subjects were asked to evaluate their pain intensity before and after each daily CES or sham treatment. Responses were scored on a scale ranging from 0 (indicating no pain) to 10 (worst possible pain).
Time Frame: Blinded Period, Unblinded Period
Population: All subjects who remained in study at each given period were analyzed. Therefore, the number of subjects examined decreased at each interval.
Measure: Mean (Standard Deviation); unit: VAS-P Score
Groups:
- Group A: BEFORE CES Treatment; Group A: AFTER CES Treatment: Subjects receiving 4 weeks of sub-sensation CES followed by 4 weeks of open label sensate treatment
- Group B: BEFORE Sham or CES Treatment; Group B: AFTER Sham or CES Treatment: Subjects receiving 4 weeks of Sham CES treatment followed by 4 weeks of open label sensate treatment
Arm/Group | Group A: BEFORE CES Treatment | Group A: AFTER CES Treatment | Group B: BEFORE Sham or CES Treatment | Group B: AFTER Sham or CES Treatment
Number analyzed (Participants) | 11 | 11 | 9 | 9
VAS-P Score
  Blinded Period: CES or Sham | 3.7 (1.7) | 3.3 (1.9) | 3.9 (1.5) | 4.2 (1.7)
  Unblinded: Open Label Sensate Period | 2.9 (2.1) | 2.3 (1.7) | 3.3 (1.4) | 2.8 (1.9)

5. Primary Outcome: Mean Visual Analogue Scale of Anxiety (VAS-A) Before and After Cranial Electrotherapy Stimulation (CES).
Description: Subjects were asked to evaluate their anxiety level before and after each daily CES treatment. Responses were scored on a scale ranging from 0 (indicating no anxiety) to 10 (worst possible).
Time Frame: Blinded Period, Unblinded Period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: VAS-A Score
Groups:
- Group B: BEFORE Treatment; Group B: AFTER Treatment: Subjects receiving 4 weeks of Sham CES treatment followed by 4 weeks of open label sensate treatment
Arm/Group | Group A: BEFORE CES Treatment | Group A: AFTER CES Treatment | Group B: BEFORE Treatment | Group B: AFTER Treatment
Number analyzed (Participants) | 11 | 11 | 9 | 9
VAS-A Score
  Blinded Period | 3.6 (2.1) | 3.2 (2.2) | 3.3 (1.7) | 3.3 (1.7)
  Unblinded, Open Label Sensate Period | 2.6 (1.9) | 2.1 (1.7) | 2.8 (1.1) | 2.3 (1.5)

6. Primary Outcome: Mean General Sleep Disturbance Scale (GSDS) Score
Description: The GSDS is a questionnaire used to qualitatively evaluate sleep. This 21-question tool evaluates each aspect of sleep and restfulness on a 0-7 score, indicating the number of days per week that each problem may be present. Total scores range from 0-147, with higher scores indicating more profound disturbances in sleep.
Time Frame: Baseline, Week 4, Week 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | A: Active/Unblinded | B: Sham/Unblinded
Number analyzed (Participants) | 11 | 9
Score
  Baseline | 76.3 (22.7) | 90.8 (13.0)
  Week 4 | 80.6 (16.4) | 83.3 (14.8)
  Week 8 | 67.8 (30.0) | 56.3 (14.6)

ADVERSE EVENTS:
Groups:
- Group A: Blinded Phase: Subjects receiving double blinded Alpha Stim 100 device preset to the lowest effective setting (1/6) for one hour daily.
- Group A: Unblinded Phase: Subjects using Alpha Stim device that has not been blinded for one hour per day for 5 days per week for 4 weeks, with settings at the patient's preference (1 to 6/6).
- Group B: Blinded Phase: Subjects receiving sham CES treatment for 1 hour daily for 4 weeks.
- Group B: Unblinded Phase: Subjects Previously receiving sham device, now using active Alpha Stim device with settings at the patient's preference (1 to 6/6), one hour per day for 5 days per week for 4 weeks.
Arm/Group | Group A: Blinded Phase | Group A: Unblinded Phase | Group B: Blinded Phase | Group B: Unblinded Phase
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/5 | 0/9 | 0/4
Other Adverse Events (participants affected / at risk) | 8/11 | 1/5 | 5/9 | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Blinded Phase (N=11) | Group A: Unblinded Phase (N=5) | Group B: Blinded Phase (N=9) | Group B: Unblinded Phase (N=4)
Ear Pain, Tingling (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Increased Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased Injury Site Pain (Nervous system disorders) | 4 (5) | 0 (0) | 2 (16) | 1 (19)
Lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night Terrors (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stiffness/ soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study had a high study turn-over rate, which led to small data group analysis. All subjects enrolled were active military service men. This made civilian and female comparison impossible. The PI also changed during study course.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes